CLINICAL TRIAL: NCT02364999
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND STUDY OF PF- 06439535 PLUS PACLITAXEL-CARBOPLATIN AND BEVACIZUMAB PLUS PACLITAXEL -CARBOPLATIN FOR THE FIRST-LINE TREATMENT OF PATIENTS WITH ADVANCED NON-SQUAMOUS NON-SMALL CELL LUNG CANCER.
Brief Title: A Comparative Study Of PF-06439535 Plus Paclitaxel-Carboplatin And Bevacizumab Plus Paclitaxel-Carboplatin Patients With Advanced Non-Squamous NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7391003; 2014-003878-16 (EudraCT Number); B7391003 (Other: Alias Study Number)
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab-Pfizer (Experimental): Bevacizumab-Pfizer plus paclitaxel and carboplatin
  Interventions: Drug: Bevacizumab-Pfizer; Drug: Paclitaxel; Drug: Carboplatin
- Bevacizumab-EU (Active Comparator): Bevacizumab-EU plus paclitaxel and carboplatin
  Interventions: Drug: Bevacizumab-EU; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab-Pfizer — Bevacizumab-Pfizer: 15 mg/kg IV on Day 1 of a 21-day cycle for each of at least 4 and no more than six (6) 21-day cycles, followed by the assigned blinded bevacizumab monotherapy.
  Arms: Bevacizumab-Pfizer
Drug: Bevacizumab-EU — bevacizumab-EU: 15 mg/kg IV on Day 1 of a 21-day cycle for each of at least 4 and no more than six (6) 21-day cycles followed by the assigned blinded bevacizumab monotherapy.
  Arms: Bevacizumab-EU
Drug: Paclitaxel — Paclitaxel 200 mg/m2 via IV infusions on Day 1 of a 21-day cycle for each of at least 4 and no more than six (6) 21-day cycles.
Drug: Carboplatin — carboplatin AUC =6.0 via IV infusions on Day 1 of a 21-day cyclefor each of at least 4 and no more than six (6) 21-day cycles.

SUMMARY:
This is a multinational, double-blind, randomized, parallel-group Phase 3 clinical trial evaluating the efficacy and safety of bevacizumab-Pfizer plus paclitaxel and carboplatin versus bevacizumab-EU plus paclitaxel and carboplatin in first-line treatment for patients with advanced (unresectable, locally advanced, recurrent or metastatic) non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age at least 18 years of age, or age of consent in the region.
* Newly diagnosed Stage IIIB or IV non-small cell lung cancer (according to Revised International System for Staging Lung Cancer criteria of 2010) or recurrent non-small cell lung cancer (NSCLC).
* Histologically or cytologically confirmed diagnosis of predominately non-squamous NSCLC.
* Be eligible to receive study treatment of bevacizumab, paclitaxel, and carboplatin based on local standard of care, for the treatment of advanced or metastatic non-squamous NSCLC.

Exclusion Criteria:

* Small cell lung cancer (SCLC) or combination SCLC and NSCLC. Squamous-cell tumors and mixed adenosquamous carcinomas of predominantly squamous nature.
* Evidence of a tumor that compresses or invades major blood vessels or tumor cavitation that is likely to bleed.
* Known sensitizing EGFR mutations (for example, deletion 19 or L858R) or EML4-ALK translocation positive mutations.
* Prior systemic therapy for NSCLC; prior neoadjuvant or adjuvant therapy is allowed if surgical resection for primary disease was performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (261):
- United States (18):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Southern Cancer Center, PC, Mobile, Alabama
  - Beaver Medical Group, L.P., Highland, California
  - Cancer Center of Central Connecticut, New Britain, Connecticut
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Swedish Covenant Hospital, Chicago, Illinois
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Holy Cross Hospital Resource Center, Silver Spring, Maryland
  - Maryland Oncology & Hematology, PA, Silver Spring, Maryland
  - Holy Cross Hospital, Hospital Pharmacy, Silver Spring, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Maryland Oncology & Hematology, PA, Wheaton, Maryland
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - Millennium Oncology, Houston, Texas
  - Millennium Oncology, Kingwood, Texas
  - Millennium Oncology, Shenandoah, Texas
  - Millennium Oncology, The Woodlands, Texas
- Australia (6):
  - Epic Pharmacy, Lismore, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Cardiac Services, John Flynn Private Hospital -, Tugun, Queensland
  - South Coast Radiology, John Flynn Private Hospital, Tugun, Queensland
  - Austin Health - Olivia Newton - John Cancer & Wellness Centre, Heidelberg, Victoria
  - Western Health, Sunshine Hospital, St Albans, Victoria
- Brazil (16):
  - Oncoclinic (Clinica de Oncologia e Atendimento de Urgencia Ltda), Fortaleza, Ceará
  - Hospital Santa Izabel / Santa Casa de Misericordia da Bahia, Salvador, Estado de Bahia
  - COT - Centro Oncologico do Triangulo Ltda, Uberlândia, Minas Gerais
  - Liga Paranaense de Combate ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Bruno Born (Sociedade Beneficencia e Caridade de Lajeado), Lajeado, Rio Grande do Sul
  - Oncosinos (Lessa Ferreira Servicos Oncologicos Ltda), Novo Hamburgo, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo - HCPF, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre - ISCMPA, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre - Hospital Santa Rita, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia - Uniao Brasileira de Educacao e Assistencia, Porto Alegre, Rio Grande do Sul
  - Instituto Joinvillense de Hematologia e Oncologia SS Ltda - Clinica de Hematologia e Oncologia, Joinville, Santa Catarina
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto -, São José do Rio Preto, São Paulo
  - Instituto de Oncologia de Sorocaba - ONCO Clinicas Especializadas SC Ltda, Sorocaba, São Paulo
  - Instituto COI de Pesquisa, Educacao e Gestao - COI Clinicas Barra Da Tijuca, Rio de Janeiro
  - lnstituto do Cancer do Estado de Sao Paulo - Octavio Frias de -, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual - IAMSPE/HSPE-FMO, São Paulo
- Complex Oncological Center Shumen EOOD, Shumen, Bulgaria
- Chile (6):
  - Instituto Clinico Oncologico del Sur (ICOS), Temuco, Región de la Araucanía
  - Instituto Clínico Oncológico del Sur (ICOS), Temuco, Región de la Araucanía
  - Centro de Investigaciones Clinicas Vina del Mar Ltda., Viña del Mar, Región de Valparaíso
  - Bradford Hill Centro de Investigaciones Clinicas, Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos (CIEC), Santiago, Santiago Metropolitan
  - Fresenius Kabi Chile, Therapia i.v., Santiago, Santiago Metropolitan
- University Hospital Centre "Sestre Milosrdnice", Zagreb, Croatia
- Czechia (5):
  - Nemocnice na Plesi s.r.o, Nová Ves pod Pleší
  - Nemocnice Novy Jicin a.s, Nový Jičín
  - Lekarna Agel Novy Jicin, Nový Jičín
  - Nemocnice Pelhrimov p.o, Radioterapeuticke oddeleni, Pelhřimov
  - Lekarna Oblastni nemocnice Pribram, Příbram
- France (4):
  - Centre Hospitalier General De Mont De Marsan, Mont-de-Marsan
  - Centre Hospitalier Montbeliard, Montbéliard
  - L'hopital prive du Confluent S.A.S., Nantes
  - Hopital d'instruction des armees Sainte Anne, Toulon
- Germany (40):
  - Klinikum Bayreuth GmbH, Bayreuth
  - Evangelische Lungenklinik Berlin, Berlin
  - Viereck-Apotheke, Berlin
  - Vivantes GmbH Apotheke des Humboldt-Klinikums, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Staedtisches Klinikum Braunschweig gGmbH Apotheke, Braunschweig
  - Staedtisches Klinikum Braunschweig gGmbH Institut fuer Roentgendiagnostik und Nuklearmedizin, Braunschweig
  - Staedtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Apotheke Johannstadt Sven Ullrich e.K., Dresden
  - Klinikum Esslingen GmbH, Esslingen a.N.
  - Radiologie Nuklearmedizin Adickesallee, Frankfurt am Main
  - St. Elisabethen - Krankenhaus, Frankfurt am Main
  - Sued-Apotheke, Frankfurt am Main
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - Johannes-Apotheke, Gröbenzell
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH - Apotheke, Halle
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH - Institut fuer Radiologie, Halle
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Zytoservice Deutschland GmbH, Hamburg
  - Katholisches Marienkrankenhaus gGmbH, Hamburg
  - Institut fuer Diagnostische und Interventionelle Radiologie, Hanover
  - Medizinische Hochschule Hannover Zentralapotheke, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum des Saarlandes - Klinik fuer Diagnostische und Interventionelle Radiologie, Homburg/Saar
  - Universitaetsklinikum des Saarlandes - Klinik fuer Innere Medizin V - Pneumologie, Allergologie,, Homburg/Saar
  - Universitaetsklinikum des Saarlandes, Apotheke, Homburg/Saar
  - Vincentius-Diakonissen-Kliniken gAG Karlsruhe, Karlsruhe
  - Vincentius-Diakonissen-Kliniken gAG Klinik fuer Diagnostische und Interventionelle Radiologie, Karlsruhe
  - Vincentius-Diakonissen-Kliniken gAG Zentralapotheke, Karlsruhe
  - Institut Fuer Versorgungsforschung In Der Onkologie, Koblenz
  - Radiologisches Institut Koblenz, Koblenz
  - Sonnenschein Apotheke, Koblenz
  - Hirsch-Apotheke, Leer
  - Onkologie UnterEms, Leer
  - Zentrum fuer Radiologie und Nuklearmedizin am Johannisplatz (ZRN Leipzig), Leipzig
  - Arkana Apotheke OHG, Leipzig
  - POIS Leipzig GbR, Pneumologisch/onkologisch/internistisches Studienzentrum, Leipzig
  - Onkologie Moers GbR, Moers
  - Friedrich-Ebert-Krankenhaus Neumuenster, Neumünster
- Greece (8):
  - University Hospital of Heraklion, Heraklion, Crete
  - Univ. of Athens Hosp. of Chest Diseases of Athens ''Sotiria'', Athens
  - General Oncology Hospital of Kifissia "Ag. Anargiroi", Athens
  - University General Hospital Of Patras, Pátrai
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - European Inter-Balkan Medical Centre, Thessaloniki
  - Thermi Clinic S.A, Thessaloniki
  - Gen.Hospital "G. Papanikolaou", Thessaloniki
- Hungary (9):
  - Semmelweis Egyetem Klinikai Pulmonologiai Klinikai Gyogyszertar, Budapest
  - Semmelweis Egyetem, Pulmonologiai Klinika, Budapest
  - Csongrad Megyei Mellkasi Betegsegek Szakkorhaza, Deszk
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű
  - Petz Aladar Megyei Oktato Korhaz, Pulmonologiai Osztaly, Győr
  - Matrai Gyogyintezet Pulmonologiai Osztaly, Mátraháza
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz - Rendelointezet, Megyei Onkologiai Kozpont, Szolnok
  - Tudogyogyintezet Torokbalint, Törökbálint
  - Zala Megyei Korhaz, Zalaegerszeg
- India (6):
  - Mahatma Gandhi Cancer Hospital And Research Institute, Visakhapatnam, Andhra Pradesh
  - HealthCare Global Enterprises Limited, Bangalore, Karnataka
  - Shatabdi Super Speciality Hospital, Nashik, Maharashtra
  - Sahyadri Clinical Research and Development Center (A Unit of Sahayadri hospitals Limited), Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Institute of Respiratory Diseases, SMS Medical College & Hospital, Jaipur, Rajasthan
- Italy (8):
  - UOC Oncologia, Treviglio, BG
  - Oncologia Medica, Fondazione Poliambulanza Instituto Ospedaliero, Brescia, BS
  - UO Oncologia Medica, Catania, CT
  - Unita di Oncologia Toracica, Meldola, FC
  - UOC di Oncologia Medica, Lido di Camaiore, LU
  - UOSD Pneumologia Oncologica - Padiglione Flaiani, Roma, RM
  - S.C. Oncologia Medica-Presidio Ospedaliero Sondrio, Sondrio, SO
  - UOC Oncologia Medica, Legnago, VR
- Japan (15):
  - National Hospital Organization Hirosaki National Hospital, Hirosaki, Aomori
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - National Hospital Organization Himeji Medical Center, Himeji, Hyōgo
  - National Hospital Organization Mito Medical Center, Higashi-ibaraki-gun, Ibaraki
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - National Hospital Organization Mie Chuo Medical Center, Tsu, Mie-ken
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - National Hospital Organization Tokyo National Hospital, Kiyose, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - National Hospital Organization Kochi National Hospital, Kochi
  - Japanese Red Cross Okayama Hospital, Okayama
  - National Hospital Organization Oita Medical Center, Ōita
- Malaysia (3):
  - Nilai Medical Centre, Kampung Baharu Nilai, Negeri Sembilan
  - Mount Miriam Cancer Hospital, Tanjung Bungah, Pulau Pinang
  - Penang Adventist Hospital, George Town
- Netherlands (4):
  - Klinisch Chemisch en Hematologisch Laboratorium (KCHL), Arnhem
  - Rijnstate Ziekenhuis, Arnhem
  - Ziekenhuis De Gelderse Vallei, Ede
  - Elkerliek Ziekenhuis, Helmond
- Philippines (2):
  - Cebu Doctors' University Hospital, Cebu City, CEBU
  - Davao Doctors Hospital, Davao City, Davao DEL SUR
- Poland (10):
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. Kopernika w Lodzi,, Lodz
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc w Olsztynie, Olsztyn
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im.Eugenii i Janusza Zeylandow, Poznan
  - MRUKMED. Lekarz Beata Madej Mruk i Partner. Sp. p. Oddzial nr 1 w Rzeszowie, Rzeszów
  - Samodzielny Publiczny Wojewodzki Szpital Zespolony w Szczecinie Szpital Wojewodzki w, Szczecin-Zdunowo
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu Szpital Obserwacyjno-Zakazny, Torun
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Wojskowy Instytut Medyczny, Klinika Onkologii, Warsaw
  - Wojewodzki Szpital Chorob Pluc im. dr Alojzego Pawelca, Wodzisław Śląski
- Romania (16):
  - SPAD Imaging International S.R.L, Craiova, Dolj
  - SC Cardio-Center SRL, Craiova, Dolj
  - SC Oncolab SRL, Oncologie, Craiova, JUD DOLJ
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Cardiologie, Târgu Mureş, Mureș County
  - Spitalul Clinic Judetean Mures, radiologie si imagistica medicala, Târgu Mureş, Mureș County
  - Spitalul Clinic Judetean Mures, sectia Clinica de Oncologie Medicala, Târgu Mureş, Mureș County
  - S.C. Oncocenter Oncologie Clinica SRL, Timișoara, Timiș County
  - Medisprof, Cluj-Napoca
  - Spitalul Clinic Municipal, Cluj-Napoca
  - SC Hiperdia SA, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta "Sf Apostol Andrei" Constanta Clinica Oncologie Medicala, Constanța
  - Centrul Medical Pozimed, SC Pozitron Medical Investigation SRL, Constanța
  - S.C. Centrul de Oncologie Sf. Nectarie S.R.L., Oncologie Medicala, Craiova
  - SC Radiotherapy Center Cluj SRL, Jud Cluj
  - Hiperdia Timisoara, Cardiologie, Timișoara
  - Hiperdia Timisoara, Radiologie si imagistica medicala, Timișoara
- Russia (32):
  - Dr's Grineva Private Clinic, Sochi, Krasnodarskiy Kray
  - SHI Oncology Dispensary #2 of Health Department of Krasnodar Region, Sochi, Krasnodarskiy Kray
  - "SAHI of Moscow ""Moscow City Oncology Hospital #62 of Health Department of Moscow""", P/o Stepanovskoe, Moscow Oblast
  - "RBHI ""Kursk Regional Clinical Oncology Dispensary"" of Healthcare Committee of Kursk Region", Kislino Steading of Kursk Region, Ryshkovskiy Village Council
  - Federal State Budgetary Institution of Healthcare "Clinical Hospital #, Lermontov, Stavropol Kray
  - SBHI of Stavropol Region "Pyatigorsk Oncology Dispensary", Pyatigorsk, Stavropol Kray
  - Stavropol Krai State Budget Healthcare Institute "Stavropol Regional Oncology Clinic", Stavropol, Stavropol Kray
  - SBHI of Stavropol Region "Essentuki Central City Hospital", Yessentuki, Stavropol Kray
  - S.G. Primushko Republican Clinical Oncology Dispensary, Izhevsk, Udmurt Republic
  - SBHI of Vladimir Region "Regional Clinical Oncology Dispensary", Vladimir, Vladimirskaya Oblast’
  - State Budget Healthcare Institution of Arkhangelsk Region, Arkhangelsk
  - Evimed Llc, Chelyabinsk
  - Chelyabinsk Regional Hospital, Chelyabinsk
  - SBHI "Chelyabinsk Regional Clinical Hospital", Chelyabinsk
  - "SBHI ""Chelyabinsk Regional Clinical Oncology Dispensary""", Chelyabinsk
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - MRT-Expert, LLC, Chelyabinsk
  - Road Clinical Hospital on the station Chelyabinsk of OJSC "RZD", Chelyabinsk
  - SBHI "Regional clinical hospital #2" of MoH of Krasnodar Region, Krasnodar
  - FSBI "N.N.Blokhin Russian Cancer Research Center" RAMS, Moscow
  - P.A.Hertsen Moscow Oncology Research Institute - Branch of the National Medical Radiological, Moscow
  - Privolzhskiy District Medical Center of Federal Biomedical Agency, Nizhny Novgorod
  - SBHI NR Clinical Diagnostic Center, Nizhny Novgorod
  - SBHI of NNR Nizhniy Novgorod Regional Oncology Dispensary, Nizhny Novgorod
  - "Budgetary Healthcare Institution of Omsk Region ""Clinical Oncology Dispensary""", Omsk
  - SBEI HPE RyazSMU of MoH of Russia based on SBI of Ryazan Region, Ryazan
  - FSBI 'Scientific-Research Oncology Institute n.a. N.N.Petrov' of MoH of RF, Saint Petersburg
  - SPb SBHI "City Clinical Oncology Dispensary", Saint Petersburg
  - Saratov scientific research institute of traumatology and orthopedics, Saratov
  - NHI Road clinical hospital at the st. Saratov II of OJSC Russian Railways, Saratov
  - Clinical hospital n.a. S.R. Mirotvortseva of SSMU, Saratov
  - Limited Liability Company "Common health", Sochi
- South Africa (5):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Amanzimtoti Oncology Centre, eManzimtoti, KwaZulu-Natal
  - Drs Schnetler, Corbett and Partners Inc, Cape Town, Western Cape
  - Dr Lior Sareli Inc, Cape Town, Western Cape
  - Cape Town Oncology Trials (Pty) Ltd, Kraaifontein, Western Cape
- South Korea (5):
  - VHS Medical Center, Seoul, Gangdong-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Spain (8):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Servicio de Oncologia, Madrid
  - Consorcio Hospital Universitario General De Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
- Changhua Christian Hospital, Changhua, Taiwan
- Thailand (8):
  - Chulalongkorn University, Patumwan, Bangkok
  - Chiangrai Prachanukroh Hospital, Muang, Changwat Chiang Rai
  - Chula Clinical Research Center, Bangkok
  - Clinical Research Center, Phramongkutklao Hospital, Bangkok
  - Medical Oncology Unit, Department of Medicine, Phramongkutklao Hospital, Bangkok
  - Division of Medical Oncology, Department of Medicine, Faculty of Medicine Siriraj Hospital,, Bangkok
  - Prachachuen Imaging Center Co., Ltd., Bangkok
  - Oncology Unit, Department of Medicine, Faculty of Medicine, Naresuan University, Phitsanulok
- Turkey (Türkiye) (14):
  - Baskent Universitesi Tip Fakultesi Adana Hastanesi, Adana
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Diskapi Yildirim Beyazit Egitim ve Arastirma Hastanesi, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Yildirim Beyazit Universitesi Tip Fakultesi Ataturk Egitim ve Arastirma Hastanesi, Ankara
  - Yedikule Gogus Hastaliklari ve Gogus Cerrahisi, Istanbul
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Onkoloji Enstitusu, Istanbul
  - Iyitem Goruntuleme ve Tani Merkezi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Ic Hastaliklari, Istanbul
  - Prof Dr Nuri Tenekeci Tani Merkezi, Istanbul
  - Euromed Goruntuleme ve Tani Merkezi, Istanbul
  - Ege Universitesi Tip Fakultesi lc Hastaliklari Anabilim Dali, Izmir
- Ukraine (10):
  - LLC "Medical clinic "INNOVACIA", chemotherapy department, Liutizh, Kyiv Oblast
  - "Municipal Institution ""Chernivtsi Regional Clinical Oncology Dispensary"",, Chernivtsi
  - MI 'City Dnipropetrovsk Multi-field Clin. Hospital #4 of DRC', Dep.-nt of Chemotherapy;, Dnipropetrovsk
  - Communal Non-Profit Enterprise "Regional Center of Oncology",, Kharkiv
  - MI 'Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council', Kryvyi Rih
  - Lviv State Oncologic Regional Treatment and Diagnostic Center, Lviv
  - Poltava Reg. Clinical Oncology Dispensary of PRC, thoracic department, SHEI of Ukr., Poltava
  - "RMI ""Sumy Reg. Clin. Oncology Dispensary"". oncothoracic dep.-nt. Surny State Univ.,, Sumy
  - "Central City Clinical Hospital, City Oncology Center, SHEI ""Uzhhorod National University"", Uzhhorod
  - Vinnytsia Regional Clinical Oncology Dispensary, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Li CSW, Sweeney K, Cronenberger C. Population pharmacokinetic modeling of PF-06439535 (a bevacizumab biosimilar) and reference bevacizumab (Avastin(R)) in patients with advanced non-squamous non-small cell lung cancer. Cancer Chemother Pharmacol. 2020 Mar;85(3):487-499. doi: 10.1007/s00280-019-03946-8. Epub 2019 Nov 26. PMID 31768697
- [Derived] Reinmuth N, Bryl M, Bondarenko I, Syrigos K, Vladimirov V, Zereu M, Bair AH, Hilton F, Liau K, Kasahara K. PF-06439535 (a Bevacizumab Biosimilar) Compared with Reference Bevacizumab (Avastin(R)), Both Plus Paclitaxel and Carboplatin, as First-Line Treatment for Advanced Non-Squamous Non-Small-Cell Lung Cancer: A Randomized, Double-Blind Study. BioDrugs. 2019 Oct;33(5):555-570. doi: 10.1007/s40259-019-00363-4. PMID 31338773
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7391003&StudyName=A%20Phase%203%20Randomized%2C%20Double-blind%20Study%20Of%20Pf%2006439535%20Plus%20Paclitaxel-carboplatin%20And%20Bevacizumab%20Plus%20Paclitaxel%20-carboplatin%20For%20The%20First-line%20Treatment%20Of%20Patients%20With%20Advanced%20Non-squamous%20Non-small%20Cell%20Lung%20Cancer.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 719 participants were enrolled in this study, and 5 of them did not receive any therapy. One (1) additional participant received only chemotherapy, and did not receive blinded bevacizumab.
Groups:
- PF-06439535: Participants received up to a maximum of 6 cycles of PF-06439535 (initial dose was 15 mg/kg) plus paclitaxel (initial dose was 200 mg/m*2) and carboplatin (initial dose was AUC 6, based on participant's pre-existing renal function and desired platelet nadir), followed by PF-06439535 monotherapy until disease progression, unacceptable toxicity, discretion of the investigator, regulatory request, death, withdrawal of consent occurred. All 3 drugs were given by intravenous (IV) infusion on Day 1 in each 21-day cycle and dose reduction was allowed for paclitaxel and carboplatin in response to toxicity. Paclitaxel was administered before carboplatin.
- Bevacizumab-EU: Participants received up to a maximum of 6 cycles of Bevacizumab-EU (initial dose was 15 mg/kg) plus paclitaxel (initial dose was 200 mg/m*2) and carboplatin (initial dose was AUC 6, based on participant's pre-existing renal function and desired platelet nadir), followed by Bevacizumab-EU monotherapy until disease progression, unacceptable toxicity, discretion of the investigator, regulatory request, death, withdrawal of consent occurred. All 3 drugs were given by intravenous (IV) infusion on Day 1 in each 21-day cycle and dose reduction was allowed for paclitaxel and carboplatin in response to toxicity. Paclitaxel was administered before carboplatin.
Period: Overall Study
Arm/Group | PF-06439535 | Bevacizumab-EU
Started | 358 | 361
Received Treatment | 356 | 358
Completed | 193 | 188
Not Completed | 165 | 173
Not completed — Death | 136 | 138
Not completed — Lost to Follow-up | 10 | 15
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 14 | 14
Not completed — Other | 0 | 1
Not completed — Randomized but did not receive treatment | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the Intent-to-Treat (ITT) population and it included all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06439535 | Bevacizumab-EU | Total
Number analyzed (Participants) | 358 | 361 | 719
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.5) | 60.9 (8.9) | 61.3 (9.2)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 19 | 17 | 36
  45-64 years | 198 | 222 | 420
  >= 65 years | 141 | 122 | 263
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 121 | 131 | 252
  Male | 237 | 230 | 467
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 319 | 319 | 638
  BLACK | 3 | 1 | 4
  ASIAN | 36 | 40 | 76
  OTHER | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Week 19
Description: ORR refers to percentage of participants who achieved complete response (CR) or partial response (PR) by Week 19 of the study in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 which was subsequently confirmed by Week 25. A participant achieved CR if both target and non-target lesions achieved CR, no new lesions; achieved PR if target lesions achieved CR or PR, non-target lesions were assessed as non-CR/non-PD (progressive disease), indeterminate or missing, and no new lesions. For target lesions, CR: complete disappearance of all target lesions except nodal disease (target nodes must decrease to normal size); PR: >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. For non-target lesions, CR: disappearance of all non-target lesions and normalization of tumor marker levels and all lymph nodes must be normal in size; non-CR/non-PD: persistence of any non-target lesions and/or tumor marker level above the normal limits.
Time Frame: 25 weeks
Population: The Intent-to-Treat (ITT) population was used for analysis of ORR, and it included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 358 | 361
percentage of participants | 45.3 [40.01 to 50.57] | 44.6 [39.40 to 49.89]
Statistical Analysis 1: Comparison: PF-06439535 vs Bevacizumab-EU; Test type: Equivalence — Calculated based on 2-sided Miettinen and Nurminen method without strata for risk difference for confirmed response. EU equivalence margins (95% CI in -13% to 13%); Risk Difference (RD) = 0.6531, 95% CI 2-sided [-6.6080 to 7.9082] — PF-06439535 vs Bevacizumab-EU
Statistical Analysis 2: Comparison: PF-06439535 vs Bevacizumab-EU; Test type: Equivalence — Calculated based on 2-sided Miettinen and Nurminen method without strata for risk ratio for confirmed response. US equivalence margins (90% CI in 0.73 to 1.37); Risk Ratio (RR) = 1.0146, 90% CI 2-sided [0.8856 to 1.1625] — PF-06439535 vs Bevacizumab-EU
Statistical Analysis 3: Comparison: PF-06439535 vs Bevacizumab-EU; Test type: Equivalence — Calculated based on 2-sided Miettinen and Nurminen method without strata for risk ratio for confirmed response. Japan equivalence margins (95% CI in 0.729 to 1.371); Risk Ratio (RR) = 1.0146, 95% CI 2-sided [0.8628 to 1.1933] — PF-06439535 vs Bevacizumab-EU

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: AE was defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of the causal relationship to study treatment. Treatment-emergent AEs (TEAEs) were defined as AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Causality to study treatment was determined by the investigator. Severity was graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 55 weeks
Population: The analysis population included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 356 | 358
Participants
  All-causality AE | 344 | 347
  All-causality SAE | 81 | 80
  Bevacizumab-related AE | 190 | 199
  Bevacizumab-related SAE | 23 | 17
  Grade 1 all-causality AE | 32 | 41
  Grade 2 all-causality AE | 141 | 134
  Grade 3 all-causality AE | 125 | 104
  Grade 4 all-causality AE | 25 | 44
  Grade 5 all-causality AE | 21 | 24

3. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory evaluation included hematology (hemoglobin, white blood cells, platelets and absolute neutrophil count), blood chemistry (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, serum or plasma creatinine, sodium, potassium, total calcium, magnesium, blood urea nitrogen or urea, and albumin ), coagulation (international normalized ratio for prothrombin time and activated partial thromboplastin time) and urinalysis (dipstick followed by a quantitative urine protein analysis for results of 2+ or greater).
Time Frame: 55 weeks
Population: The analysis population included all participants who were randomized and received at least 1 dose of study treatment, and had laboratory evaluation done.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 342 | 348
Participants | 303 | 304

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of PD or to death due to any cause in the absence of documented PD. DOR was based on the Brookmeyer and Crowley method.
Time Frame: 55 weeks
Population: The analysis population included participants in ITT population (all participants who were randomized to study treatment) who had a confirmed objective response achieved by Week 19.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 162 | 161
weeks | 36.3 [31.6 to 43.6] | 28.7 [27.0 to 36.3]
Statistical Analysis 1: Comparison: PF-06439535 vs Bevacizumab-EU; Test type: Other — Hazard ratio of PF-06439535 versus Bevacizumab-EU; a hazard ratio =1 indicated no difference in progressive disease(PD)/death between 2 reporting groups; >1 indicated an increase in PD/death in PF-06439535; <1 indicated an increase in PD/death in bevacizumab-EU; p = 0.1077, Log Rank; Stratified by smoking, sex and region; Hazard Ratio (HR) = 0.800, 95% CI 2-sided [0.608 to 1.051]

5. Secondary Outcome: Progression Free Survival Rate at 55 Weeks
Description: This outcome measure refers to the possibility of being progression free at 55 weeks since start of study treatment, estimated from the Kaplan-Meier curve using the product-limit method.
Time Frame: 55 weeks
Population: The ITT population was used for analysis, and it included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 358 | 361
percentage of participants | 32.3 [26.9 to 37.8] | 30.5 [25.3 to 35.8]
Statistical Analysis 1: Comparison: PF-06439535 vs Bevacizumab-EU; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.4492, Log Rank; Stratified by smoking, sex and region; Hazard Ratio (HR) = 0.931, 95% CI [0.777 to 1.116]

6. Secondary Outcome: Survival Rate at 55 Weeks
Description: This outcome measure refers to the possibility of being alive at 55 weeks since start of study treatment, estimated from the Kaplan-Meier curve using the product-limit method.
Time Frame: 55 weeks
Population: The ITT population was used for analysis, and it included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 358 | 361
percentage of participants | 65.8 [60.5 to 70.6] | 64.1 [58.6 to 69.0]
Statistical Analysis 1: Comparison: PF-06439535 vs Bevacizumab-EU; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.4726, Log Rank; Stratified by smoking, sex and region; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.729 to 1.157]

7. Secondary Outcome: Serum Concentration of Bevacizumab up to 1 Year
Time Frame: Pre-dose from Cycle 1 to Cycle 17, 2.5 hours post-dose in Cycle 1, and 1.5 hours post-dose in Cycle 5
Population: The analysis population included all participants in the per-protocol population (all participants who were randomized and received study treatment as planned and had no major protocol deviations) who had at least 1 drug concentration measurement after administration of study treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 351 | 354
ng/mL
  Pre-dose in Cycle 1: number analyzed (Participants) | 333 | 338
  Pre-dose in Cycle 1 | 68.08 (705.53) | 116.4 (1032.1)
  2.5 hours post-dose in Cycle 1: number analyzed (Participants) | 319 | 326
  2.5 hours post-dose in Cycle 1 | 280000 (103260) | 302200 (100360)
  Pre-dose in Cycle 2: number analyzed (Participants) | 310 | 326
  Pre-dose in Cycle 2 | 54350 (44479) | 58930 (49452)
  Pre-dose in Cycle 3: number analyzed (Participants) | 206 | 211
  Pre-dose in Cycle 3 | 81090 (48671) | 83350 (32384)
  Pre-dose in Cycle 4: number analyzed (Participants) | 277 | 299
  Pre-dose in Cycle 4 | 100900 (54979) | 99750 (50531)
  Pre-dose in Cycle 5: number analyzed (Participants) | 257 | 271
  Pre-dose in Cycle 5 | 105300 (48469) | 110000 (65416)
  1.5 hours post-dose in Cycle 5: number analyzed (Participants) | 192 | 201
  1.5 hours post-dose in Cycle 5 | 360700 (131170) | 377200 (142250)
  Pre-dose in Cycle 6: number analyzed (Participants) | 244 | 268
  Pre-dose in Cycle 6 | 112000 (40825) | 116700 (53844)
  Pre-dose in Cycle 7: number analyzed (Participants) | 192 | 214
  Pre-dose in Cycle 7 | 117300 (53844) | 122100 (47793)
  Pre-dose in Cycle 8: number analyzed (Participants) | 195 | 208
  Pre-dose in Cycle 8 | 123600 (48893) | 126400 (52985)
  Pre-dose in Cycle 9: number analyzed (Participants) | 184 | 193
  Pre-dose in Cycle 9 | 127200 (46200) | 140900 (62548)
  Pre-dose in Cycle 10: number analyzed (Participants) | 170 | 179
  Pre-dose in Cycle 10 | 125700 (50769) | 135900 (53975)
  Pre-dose in Cycle 11: number analyzed (Participants) | 170 | 169
  Pre-dose in Cycle 11 | 129500 (61329) | 135600 (54531)
  Pre-dose in Cycle 12: number analyzed (Participants) | 141 | 138
  Pre-dose in Cycle 12 | 135200 (64560) | 136300 (51312)
  Pre-dose in Cycle 13: number analyzed (Participants) | 136 | 121
  Pre-dose in Cycle 13 | 130900 (58093) | 139700 (53750)
  Pre-dose in Cycle 14: number analyzed (Participants) | 131 | 117
  Pre-dose in Cycle 14 | 128000 (50840) | 136200 (53439)
  Pre-dose in Cycle 15: number analyzed (Participants) | 103 | 104
  Pre-dose in Cycle 15 | 134000 (55933) | 134000 (49663)
  Pre-dose in Cycle 16: number analyzed (Participants) | 92 | 95
  Pre-dose in Cycle 16 | 137000 (54813) | 128600 (49742)
  Pre-dose in Cycle 17: number analyzed (Participants) | 90 | 92
  Pre-dose in Cycle 17 | 134800 (86847) | 127500 (52784)

8. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: ADA assay was performed using a sensitive, specific, and semi-quantitative electrochemiluminescent (ECL) method, which used biotinylated- and ruthenium-labeled PF-06439535 as reagents. Samples with ADA titer greater than or equal to (>=) 2.29 were considered positive.
Time Frame: 55 weeks
Population: The analysis population included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 356 | 358
Participants
  Cycle 1 pre-dose: number analyzed (Participants) | 351 | 353
  Cycle 1 pre-dose | 1 | 3
  Overall (post-treatment): number analyzed (Participants) | 339 | 350
  Overall (post-treatment) | 5 | 5

9. Secondary Outcome: Number of Participants With Neutralizing Antibody (NAb)
Description: Only samples that were confirmed positive for ADA were further tested for NAb. The NAb analysis was conducted using a single validated quasi-quantitative enzyme-linked immunosorbent assay (ELISA) that utilized PF-06439535 as a reagent. Samples with NAb titer >=1.70 were considered positive.
Time Frame: 55 weeks
Population: The analysis population included all participants who had positive ADA results at any time point.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06439535 | Bevacizumab-EU
Number analyzed (Participants) | 6 | 7
Participants
  Cycle 1 pre-dose: number analyzed (Participants) | 1 | 3
  Cycle 1 pre-dose | 1 | 0
  Overall (post-treatment): number analyzed (Participants) | 5 | 5
  Overall (post-treatment) | 0 | 3

ADVERSE EVENTS:
Time Frame: 55 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Groups:
- Total: This reporting group include all participants who received at least 1 dose of study treatment from PF-06439535 and Bevacizumab-EU groups.
Arm/Group | PF-06439535 | Bevacizumab-EU | Total
All-Cause Mortality (participants affected / at risk) | 144/356 | 149/358 | 293/714
Serious Adverse Events (participants affected / at risk) | 81/356 | 80/358 | 161/714
Other Adverse Events (participants affected / at risk) | 328/356 | 333/358 | 661/714
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06439535 (N=356) | Bevacizumab-EU (N=358) | Total (N=714)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 5 (6) | 7 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (7) | 7 (7) | 12 (14)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 6 (8) | 10 (13)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5) | 3 (3) | 6 (8)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (3) | 4 (6)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Asthenia (General disorders) | 4 (5) | 1 (1) | 5 (6)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Death (General disorders) | 2 (2) | 3 (3) | 5 (5)
Disease progression (General disorders) | 4 (4) | 5 (5) | 9 (9)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1) | 3 (3)
Cholangitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 8 (11) | 6 (6) | 14 (17)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3) | 3 (4)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2) | 4 (5)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 3 (4) | 3 (4)
Mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2) | 9 (9)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Brachiocephalic vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Subgaleal haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06439535 (N=356) | Bevacizumab-EU (N=358) | Total (N=714)
Leukopenia (Blood and lymphatic system disorders) | 26 (44) | 30 (56) | 56 (100)
Neutropenia (Blood and lymphatic system disorders) | 59 (130) | 66 (144) | 125 (274)
Thrombocytopenia (Blood and lymphatic system disorders) | 55 (122) | 66 (125) | 121 (247)
Constipation (Gastrointestinal disorders) | 39 (45) | 27 (36) | 66 (81)
Diarrhoea (Gastrointestinal disorders) | 46 (59) | 48 (66) | 94 (125)
Nausea (Gastrointestinal disorders) | 71 (111) | 69 (112) | 140 (223)
Vomiting (Gastrointestinal disorders) | 41 (52) | 33 (42) | 74 (94)
Asthenia (General disorders) | 46 (78) | 43 (65) | 89 (143)
Fatigue (General disorders) | 73 (110) | 71 (87) | 144 (197)
Pyrexia (General disorders) | 24 (31) | 23 (41) | 47 (72)
Infusion related reaction (Injury, poisoning and procedural complications) | 19 (26) | 22 (26) | 41 (52)
Alanine aminotransferase increased (Investigations) | 49 (95) | 39 (53) | 88 (148)
Aspartate aminotransferase increased (Investigations) | 44 (94) | 37 (59) | 81 (153)
Blood alkaline phosphatase increased (Investigations) | 29 (46) | 32 (48) | 61 (94)
Blood creatinine increased (Investigations) | 16 (28) | 21 (33) | 37 (61)
Platelet count decreased (Investigations) | 23 (31) | 19 (38) | 42 (69)
Weight decreased (Investigations) | 36 (43) | 29 (40) | 65 (83)
Decreased appetite (Metabolism and nutrition disorders) | 48 (76) | 46 (65) | 94 (141)
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 (82) | 43 (71) | 83 (153)
Bone pain (Musculoskeletal and connective tissue disorders) | 25 (58) | 23 (47) | 48 (105)
Myalgia (Musculoskeletal and connective tissue disorders) | 54 (131) | 49 (109) | 103 (240)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (23) | 23 (29) | 39 (52)
Headache (Nervous system disorders) | 30 (35) | 37 (45) | 67 (80)
Neuropathy peripheral (Nervous system disorders) | 53 (67) | 65 (86) | 118 (153)
Paraesthesia (Nervous system disorders) | 40 (64) | 31 (36) | 71 (100)
Peripheral sensory neuropathy (Nervous system disorders) | 34 (45) | 46 (70) | 80 (115)
Polyneuropathy (Nervous system disorders) | 23 (34) | 19 (22) | 42 (56)
Proteinuria (Renal and urinary disorders) | 28 (50) | 34 (76) | 62 (126)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (53) | 47 (58) | 88 (111)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 (38) | 35 (41) | 67 (79)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 40 (51) | 32 (48) | 72 (99)
Alopecia (Skin and subcutaneous tissue disorders) | 166 (216) | 165 (232) | 331 (448)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 21 (29) | 30 (39)
Hypertension (Vascular disorders) | 60 (83) | 62 (110) | 122 (193)
Anaemia (Blood and lymphatic system disorders) | 102 (196) | 106 (200) | 208 (396)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT02364999/SAP_000.pdf
  • Study Protocol (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT02364999/Prot_001.pdf